CLINICAL TRIAL: NCT03421171
Title: Ethical Dilemmas in Anaesthesiology in the Netherlands; a Qualitative Interview Study.
Acronym: AnaesthEthics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, E.A. Kwofie, doctoranda, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: AE1-AMC
Record Dates: First submitted 2018-01-23; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Ethical Dilemmas; Ethical Issues; Moral Issues; Moral Dilemmas; Anaesthesiology; Anaesthesiologist

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — Qualitative research through semi-structured interviews

SUMMARY:
This study will describe which ethical dilemmas are experienced by anesthesiologist in the Dutch Healthcare system and what the current solving strategies are for these issues. Semi- structured interviews will be conducted with anaesthesiologists employed in different hospitals in the Netherlands..

DETAILED DESCRIPTION:
Ethical considerations are part of a doctors daily practice. The development of anaesthesiologists as ' perioperative' doctors is increasingly giving anaesthesiologists a treatment function. As the third largest medical specialty, they are also involved in ethical dilemmas. Examples of common themes in the literature include:' informed consent' and professionalism. Nevertheless, good research into ethical dilemmas in the field of anaesthesiology is lacking.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Employed as anaesthesiologist
* Employed in an academic or non-academic hospital in the Netherlands

Exclusion Criteria:

* Other medical specialists
* language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: anaesthetist employed in the Netherlands working in a academic of non-academic hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-01-20 (Actual); Primary Completion 2018-12-20 (Estimated); Study Completion 2019-01-20 (Estimated)

PRIMARY OUTCOMES:
interviews (qualitative interview study) | 10 years (depends on working experience of the respondent)
  Categories of ethical dilemmas experienced during work as assessed by interviews

CONTACTS AND LOCATIONS:
Overall Officials: M. W Hollmann, Principal Investigator — AIDS Malignancy Consortium
Locations (1):
- Academic Medical Centre, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
De identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: within 6 months of study completion
Access Criteria: data acces will be reviewed. requestors will be required to sign a data access agreement